CLINICAL TRIAL: NCT06262984
Title: The Effect of the Therapeutic Play Applied Before Nasopharyngeal Swaping on Children's Emotional Manifestation in the 3-6 Years Old Group
Brief Title: Therapeutic Play Before Nasopharyngeal Swabbing in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Zeynep Erkut, Assist. Prof., Maltepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/21-754
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Behavior, Coping
Keywords: Child; Nasopharyngeal swab; Therapeutic play; Emotional manifestation
MeSH Terms: conditions — Behavior | interventions — Play Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Play Group (Experimental): The researcher will demonstrate the nasopharyngeal swabbing process on the doll with the children who have chosen a therapeutic play group, using a therapeutic play method, and play with the child. The Children's Emotional Manifestation Scale (CEMS) will be evaluated and scored by the researcher and the observing nurse.
  Interventions: Other: Therapeutic Play
- Control Group (No Intervention): Children who choose the control group will be explained the nasopharyngeal swab procedure as routinely performed in the outpatient clinic.The Children's Emotional Manifestation Scale (CEMS) will be evaluated and scored by the researcher and the observing nurse.

INTERVENTIONS:
Other: Therapeutic Play — The researcher will demonstrate the nasopharyngeal swabbing process on the doll with the children who have chosen a therapeutic play group, using a therapeutic play method, and play with the child. The Children's Emotional Manifestation Scale (CEMS) will be evaluated and scored by the researcher and the observing nurse.
  Arms: Therapeutic Play Group

SUMMARY:
The study will be conducted with the randomized controlled experimental method. Children who apply to the Child Health and Diseases Polyclinic and Child Health and Diseases Service and who will have nasopharyngeal swab applied will be divided into two groups by drawing lots. After the randomization children in the therapeutic play group the nasal swab will be shown on the doll to the child by the researcher before being taken. The child is then allowed to play with the doll accompanied by the researcher. No intervention will be performed on children in the control group. The parents will also be found next to their children in both groups during the procedure.

DETAILED DESCRIPTION:
Many different non-pharmacological methods are used to cope with negative emotional responses such as pain, stress, fear and anxiety caused by diagnostic procedures in children. One of these non-pharmacological methods is therapeutic play. Therapeutic play method applied in line with the philosophy of atraumatic care in preparation for medical diagnostic procedures can ensure children's adaptation to the procedures by reducing the negative emotional effects of these procedures on the child. Energy Expenditure Play, Dramatic Play and Creative Play are used as therapeutic play types.

The aim of this study is to determine the effect of therapeutic play applied before the nasopharyngeal swab procedure on the emotional indicators of children aged 3-6 years who apply to the pediatric clinic and pediatric service. In line with the results obtained from studies using a similar research method, the sample size of the study was determined by power analysis (G*Power 3.1.9.4). The sample size was found to be 68 children in total, with a minimum of 34 children for each group. To collect data, an information form and the Children's Emotional Manifestation Scale (CEMS) will be used. Children and their parents who apply to the pediatric service and pediatric outpatient clinic will be informed about the study. The children and parents included in the study will be informed about the research by the researcher through a face-to-face meeting, and a consent form and information form will be filled out. Children will determine their groups by drawing lots. The researcher will demonstrate the nasopharyngeal swabbing process on the doll with the children who have chosen a therapeutic play group, using a therapeutic play method, and play with the child. Children who choose the control group will be explained the nasopharyngeal swab procedure as routinely performed in the outpatient clinic. The Children's Emotional Manifestation Scale (CEMS) will be evaluated and scored by the researcher and the observing nurse.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 3 and 6,
* Children who have not received medical attention in the last 24 hours,
* Children without speech, hearing, psychological or neurological problems,
* Children who can speak and understand Turkish at native level,
* Children and their parents who agree to participate in the research.

Exclusion Criteria:

* Being younger than 3 years old and older than 6 years old,
* Children who received medical intervention in the last 24 hours,
* Children with any speech, hearing, psychological or neurological problems,
* Children who do not speak Turkish as their native language,
* Children and their parents who do not agree to participate in the research.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Children's emotional manifestation | one minute before nasopharyngeal swabbing, when nasopharyngeal swabbing begins, one minute after nasopharyngeal swabbing
  The child's emotional response will be evaluated with the Children's Emotional Manifestation Scale (CEMS) by the researcher and the observing nurse before, during and after the procedure.
  In the scale, emotional indicators are evaluated according to 5 parameters (facial expression, voice, activity, interaction, cooperation level). These five parameters are scored from 1 to 5, with the lowest score being '5' and the highest being '25'. A higher scale score indicates that the child showed more negative emotional behavior during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Erkut, PhD, Principal Investigator — Maltepe University; Melisa Şengül, Principal Investigator — Acıbadem Hospital
Locations (1):
- Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No